# Comprehensive Assessment of Rosacea Patients' Clinical Trial Experiences: A Medical Investigation

Informed Consent Form for Rosacea Patients in <a href="Power Clinical Trial's">Power Clinical</a>
<a href="Trial's">Trial's</a> Medical Study

Date: February 17, 2023

#### About This Informed Consent Form

Power Clinical Trials is conducting an observational clinical trial, and we are inviting you to participate. We have prepared this document to provide you with a comprehensive understanding of the study and to obtain your informed consent. We encourage you to read this document carefully and to ask any questions that you may have before deciding to participate.

#### Rosacea Clinical Trial Overview

The purpose of this study is to observe patients with rosacea who are currently participating in an active interventional clinical trial. This study is important because it will help us gather important data on the condition and any associated patterns that may affect the enrolment and withdrawal rate of the participants. The information gathered from this can contribute to the advancement of medical knowledge and the development of better treatments for rosacea patients.

## What is the Study Procedure?

As a participant in this study, you will not receive any specific treatment or intervention beyond what is currently prescribed by your healthcare provider. Your medical information and health outcomes will be observed and recorded by study personnel over a period of time.

This observational study is seeking to gather additional data from participants engaged in interventional clinical trials by conducting bi-weekly surveys and quarterly check-in calls.

It is important to understand that the interventional clinical trial you are participating in is entirely separate from this observational study, and your treatment plan will not be altered in any way by participating in this study.

If you have any questions about your current interventional clinical trial, please reach out to your care team. They will be able to provide you with the information you need and address any concerns you may have.

#### Are There Risks and Benefits?

We have found no known risks associated with participating in this observational study. We aim to collect valuable data that can contribute to the advancement of medical knowledge and ultimately lead to the development of better treatments for the medical condition being studied. Please also note that participation in this study does not guarantee any personal benefits or treatment for your medical condition.

# Is My Information Safe?

All of your personal information and medical data will be kept confidential and only accessible to study personnel. Your name and other identifying information will be kept confidential and not disclosed in any reports or publications. However, it is important to note that the data collected in this study

### How Does This Trial Compare to Other Rosacea Clinical Trials?

There are several studies available to patients with various rosacea, many of which are interventional and require a specified course of therapy. However, this particular clinical trial is an observational experiment that does not require patients to participate in any specific therapy or treatment.

It is important to note that our team may not be familiar with all the available clinical trials for patients with rosacea. If you are interested in learning about other <u>rosacea studies</u>, we recommend checking out resources such as clinicaltrials.gov or Power's participant reference site, where you can find information on additional <u>rosacea clinical trials</u>.

#### Can I Read More Studies About Clinical Trial Representation?

If you want to read more on studies about clinical trial representation, here are some published works you can check:

Melloni, Chiara, Jeffrey S. Berger, Tracy Y. Wang, Funda Gunes, Amanda Stebbins, Karen S. Pieper, Rowena J. Dolor, Pamela S. Douglas, Daniel B. Mark, and L. Kristin Newby. "Representation of women in randomized clinical trials of cardiovascular disease prevention." *Circulation: Cardiovascular Quality and Outcomes* 3, no. 2 (2010): 135-142.

Denby, Kara J., Natalie Szpakowski, Julie Silver, Mary Norine Walsh, Steve Nissen, and Leslie Cho. "Representation of women in cardiovascular clinical trial leadership." *JAMA Internal Medicine* 180, no. 10 (2020): 1382-1383.

## Participant Statement

After reviewing the above material, I have had the opportunity to ask questions, and all my inquiries have been thoroughly addressed. I understand that my participation in this research study is entirely voluntary, and I may withdraw from the study at any time without penalty or consequence.

I am aware that signing this form does not waive any of my legal rights. I will receive a copy of this consent form for my records. By signing below, I am consenting to participate in this research study and agree to comply with the study's protocols and requirements to the best of my ability.

I appreciate the efforts of the research team to inform me about the study, including the purpose, procedures, potential risks, and benefits. I believe that my participation in this study could make a valuable contribution to advancing medical knowledge and improving patient care. I am committed to upholding my responsibilities as a study participant and will inform the research team of any changes to my health or status that may affect my participation in the study.

| Printed Name of Participant | |
|---|---|
| Participant Signature | |
| Date | |
| Statement of Person Getting Conse | nt |
| • | ment with the participant, I am confident that ks, benefits, alternatives, and procedures |
| Printed Name of Person Conducting In | formed Consent Discussion |
| Person Conducting Informed Consent | Discussion Signature |
| <br>Date | |